CLINICAL TRIAL: NCT03499171
Title: A Placebo-controlled Trial With Citalopram for the Treatment of Typical Reflux Symptoms in Patients With Reflux Hypersensitivity or Functional Heartburn With Incomplete Proton Pump Inhibitor Response
Brief Title: Citalopram for Reflux Hypersensitivity and Functional Heartburn
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S61111
Record Dates: First submitted 2018-04-11; First posted 2018-04-17 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citalopram (Experimental): 20mg, once a day
  Interventions: Drug: Citalopram 20mg
- Placebo (Placebo Comparator): Once a day
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Citalopram 20mg — Citalopram is taken once a day as an add-on to PPI treatment (2x/d).
  Arms: Citalopram
Drug: Placebo Oral Tablet — Placebo is taken once a day as an add-on to PPI treatment (2x/d)
  Arms: Placebo

SUMMARY:
Citalopram is a drug used in the treatment of depressive episodes and belongs to the group of selective serotonin reuptake inhibitors (SSRI). Serotonin is an important neurotransmitter predominantly found in the brain and the gastrointestinal tract. Serotonin is associated with psychological disorders, including anxiety and depression, and emotion regulation and it has been shown that anxiety and depression are associated with increased severity of GERD-related symptoms. Citalopram and other SSRI's elevate the concentration of serotonin by blocking the reabsorption into the presynaptic neuron and thereby increasing the level of serotonin available to bind the postsynaptic receptor. A recent study showed beneficial effects of citalopram in patients with reflux hypersensitivity. However, there was no objective measurement for reflux nor esophageal sensitivity during the treatment period. Moreover, the effect of citalopram in patients with functional heartburn has not been studied so far. Therefore, the inevestigators will conduct a randomized, parallel, placebo-controlled study to evaluate the efficacy of citalopram on the improvement in symptom severity, reflux parameters and esophageal sensitivity. 50 patients with reflux hypersensitivity and 50 patients with functional heartburn will receive either placebo or citalopram (Cipramil®) 20 mg as an add-on for a period of 8 weeks. Symptom severity will be assessed by a validated reflux questionnaire (ReQuest questionnaire and diaries), reflux parameters by performing a 24 hour impedance-pH monitoring and esophageal sensitivity using the multimodal esophageal stimulation paradigm

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old.
2. History of typical GERD symptoms during PPI treatment, at least 3 times per week for 12 weeks.
3. Daily intake of PPI treatment 12 weeks prior to inclusion, with at least 8 weeks of b.i.d. therapy (at least 2*20mg of omeprazole or equivalent).
4. Sexually active women of child bearing potential participating in the study must use a medically acceptable form of contraception. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception.
5. Subjects must be capable of understanding and be willing to provide signed and dated written voluntary informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

1. Endoscopic signs of severe erosive esophagitis (≥ grade B, Los Angeles classification) on endoscopy performed during PPI treatment in the 6 months prior to screening.
2. Systemic diseases, known to affect esophageal motility.
3. Surgery in the thorax or in the upper part of the abdomen (appendectomy and cholecystectomy are allowed).
4. QT c>450 ms
5. Treatment with SSRI's prior to the start of the study.
6. Concomitant use of medications such as: anticholinergics, tricycle antidepressants, baclofen and prokinetics.
7. Significant neurological, respiratory, hepatic, renal, hematological, cardiovascular, metabolic or gastrointestinal cerebrovascular disease as judged by the investigator.
8. Major psychiatric disorder.
9. Absence of PPI intake for at least 2 consecutive days in the 2 weeks prior to the screening.
10. Pregnancy or breast feeding.
11. History of poor compliance. History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent.
12. History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
change in number of reflux episodes | 8 weeks
  The primary efficacy endpoint will be the change in number of reflux episodes assessed by 24 hour impedance-pH monitoring.

SECONDARY OUTCOMES:
change in reflux parameters | 8 weeks
  change in reflux parameters (number of reflux episodes with a high proximal extent, volume exposure) assessed by 24 hour impedance-pH monitoring,
change in esophageal sensitivity | 8 weeks
  change in esophageal sensitivity assessed by multimodal esophageal stimulation procedure
change in symptom severity | 8 weeks
  change in symptom severity assessed by validated reflux questionnaires (ReQuest questionnaire and diaries). Patients will have to indicate the symptom occurence and symptom severity on a scale. Two words, on each site of the scale indicate their symptom severity (on the left "totally not present" on the right "very strong present"). A higher score represents a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No